CLINICAL TRIAL: NCT04007614
Title: Bone Health in Adolescents and Young Adults With Oral Macro-progestin Treatment : Observational Study
Brief Title: Bone Health in Adolescents and Young Adults With Oral Macro-progestin Treatment
Acronym: MACROS
Status: Withdrawn | Type: Observational
Why Stopped: The study never started
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190093; IDRCB : 2019-A00340-57 (Other: ANSM)
Record Dates: First submitted 2019-04-17; First posted 2019-07-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2022-11

CONDITIONS: Contraception; Macro-progestins
Keywords: Macro-progestins; Bone health
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients who have taken a macro progestin treatment for more than 6 months between 16 and 25 years of age.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Fardellone questionnaire (evaluation of calcium intake) Tolerance of treatment

SUMMARY:
Many factors are known to influence the acquisition of bone capital, especially estrogens in women. Estrogens have a major role in bone growth and the acquisition of bone mass peaks during puberty. This peak of bone mass is an important determinant of the risk of osteoporotic fracture in adulthood.

It is known that estrogen deficiency increases the rate of bone remodeling and engenders an imbalance between resorption and bone formation, which can lead to osteoporosis.

Oral estroprogestin contraceptives have an anti-gonadotropic effect and suppress estrogen secretion by the ovaries.

However, studies in adolescents and young adults are rare and evidence of an effect on bone is still inconclusive, although there is increasing evidence that oral estroprogestin contraceptives in teenage girls may compromise the performance of the bone mass.

Macro progestins treatments are prescribed in France to patients with contraindications to estroprogestin treatments. This practice is french and few recommendations exist on the use of these molecules by the oral route. There are no studies that describe the impact of these oral treatments on the bone health of young women treated.

The Department of endocrinology, gynecology and pediatric diabetes of Necker-Enfants Malades hospital, follows many young girls taking a macro progestin treatment. This study is exclusively descriptive and will focus on the clinical and medical datas available on the bone health of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 to 25 years old
* Patients followed at Necker-Enfants Malades hospital
* Patients who have taken or taking macro-progestins treatment by oral route (Luteran, Lutenyl, Surgestone) for at least 6 months between the age of 16 and 25 years

Exclusion Criteria:

* Patients with a pathology or treatment that can alter bone mineral density

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Macroprogestins treatment.
Study Population: Patients followed by the department of endocrinology, gynecology and pediatric diabetes of Necker hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Bone densitometry | Day 0
  Z score values compared to the reference values
Calcemia | Day 0
  Blood test
Ionized calcium | Day 0
  Blood test
Phosphor | Day 0
  Blood test
Magnesium | Day 0
  Blood test
Albumin | Day 0
  Blood test
Parathormone | Day 0
  Blood test
25 OH vitamin D3 | Day 0
  Blood test
Creatinine | Day 0
  Blood test
Osteocalcin | Day 0
  Blood test
Bone alkaline phosphatase isoenzymes | Day 0
  Blood test
C-terminal telopeptide of type I collagen | Day 0
  Blood test
Calciuria | Day 0
  Urine test
Natriuresis | Day 0
  Urine test
Creatinuria | Day 0
  Urine test

SECONDARY OUTCOMES:
Clinical tolerance of treatment | Day 0
  6 questions asked to the patient under treatment, a yes or no answer is expected : presence of menstruating, regularity of cycles, out-of-periods bleeding, weight gain, acne, satisfaction in relation to treatment.
Follicle stimulating hormone | Day 0
  Blood test, patients under macro progestin treatment at day 0
Gonadotrophin b LH | Day 0
  Blood test, patients under macro progestin treatment at day 0
Estradiol | Day 0
  Blood test, patients under macro progestin treatment at day 0

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Da Costa, MD, Study Director — Hôpital Necker-Enfants Malades
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, Paris, France